CLINICAL TRIAL: NCT05111496
Title: Evaluation of the Radiological Dose Delivered to Risky Interventional Cardiology Patients (Optidose)
Acronym: Optidose
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Collaborators: European Clinical Trial Experts Network (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-A02398-49
Record Dates: First submitted 2021-10-27; First posted 2021-11-08 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-10

CONDITIONS: X-rays; Effects; Chronic Total Occlusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient requiring intervention (complex coronary dilation or coronary recanalization): Patient requiring intervention with a predicted risk of exceeding the radiological threshold (Air Kerma> 3Gy): complex coronary dilation, coronary recanalization
  Interventions: Radiation: Gafchromic film

INTERVENTIONS:
Radiation: Gafchromic film — Before the X-ray radiation, a Gafchromic film will be placed on the patient's back at the start of the operation

SUMMARY:
The purpose of this study is therefore to study the actual doses of X-rays delivered to the patient's skin during recanalization of a coronary artery in a context of Chronic Total Occlusion

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years-old
* Patient requiring intervention with a predicted risk of exceeding the radiological threshold (Air Kerma> 3Gy): complex coronary dilation, coronary recanalization
* Patient benefiting from a social protection insurance
* Patient having been informed and not objecting to this research

Exclusion Criteria:

* Patient refusal to participate in the study
* Patient with known radiosensitivity factors (eg: Lupus)
* Patient having had radiotherapy treatment of the thoracic region.
* Patient whose sum of radiation doses to the skin> 0.5 Gy in the thoracic region in the 3 months preceding inclusion.
* Patient participating in another clinical study
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision
* Pregnant or breastfeeding woman
* Patient hospitalized without consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient over 18 years-old, requiring intervention with a predicted risk of exceeding the radiological threshold (Air Kerma> 3Gy): complex coronary dilation, coronary recanalization
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2020-09-24 (Actual); Primary Completion 2021-10-06 (Actual); Study Completion 2021-11-24 (Estimated)

PRIMARY OUTCOMES:
Dose measured to the patient's skin at the entrance to the X-ray beam | 1 month
  Dose expressed in Gy (Peak skin dose).

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital privé La Louvière, Lille, Haut de France, France